CLINICAL TRIAL: NCT03027154
Title: For Tuberculosis (TB) Clinical Auxiliary Diagnosis of Recombinant Mycobacterium Tuberculosis Allergen ESAT6-CFP10 Dose Certain Phase III Clinical Research in Children Under the Age of 18 Years Old
Brief Title: Clinical Study of Recombinant Mycobacterium Tuberculosis ESAT6-CFP10 Allergen for Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government); Beijing Children's Hospital (Other); Wuhan Institute for Tuberculosis Control (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: LTao-EC III-children
Record Dates: First submitted 2017-01-19; First posted 2017-01-23 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2017-10

CONDITIONS: Tuberculosis Diagnosis
Keywords: diagnostic test; children; diagnosis of tuberculosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TB subjects in 5-18 years old (Experimental): 24 cases TB subjects in 5-18 years old are injected ESAT6-CFP10 in left arm and TB-PPD in right arm or ESAT6-CFP10 in right arm and TB-PPD in left arm. For each of participant,the person in this clinical research, the study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h.
  Interventions: Biological: ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: ESAT6-CFP10 in right arm and TB-PPD in left arm
- non-TB subjects in 5-18 years old (Experimental): 24 cases non-TB subjects in 5-18 years old are injected ESAT6-CFP10 in left arm and TB-PPD in right arm or ESAT6-CFP10 in right arm and TB-PPD in left arm. For each of participant,the person in this clinical research, the study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h.
  Interventions: Biological: ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: ESAT6-CFP10 in right arm and TB-PPD in left arm
- TB subjects under 5 years old (Experimental): 24 cases TB subjects under 5 years old are injected ESAT6-CFP10 in left arm and TB-PPD in right arm or ESAT6-CFP10 in right arm and TB-PPD in left arm. For each of participant,the person in this clinical research, the study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h.
  Interventions: Biological: ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: ESAT6-CFP10 in right arm and TB-PPD in left arm
- non-TB subjects under 5 years old (Experimental): 24 cases non-TB subjects under 5 years old are injected ESAT6-CFP10 in left arm and TB-PPD in right arm or ESAT6-CFP10 in right arm and TB-PPD in left arm. For each of participant,the person in this clinical research, the study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h.
  Interventions: Biological: ESAT6-CFP10 in left arm and TB-PPD in right arm; Biological: ESAT6-CFP10 in right arm and TB-PPD in left arm

INTERVENTIONS:
Biological: ESAT6-CFP10 in left arm and TB-PPD in right arm — All subjects including TB subjects in 5-18 years old、non-TB subjects in 5-18 years old、TB subjects under 5 years old and non-TB subjects under 5 years old inject ESAT6-CFP10 in left arm and TB-PPD in right arm respectively. Two drug must use at the same participant and in different arms.
Biological: ESAT6-CFP10 in right arm and TB-PPD in left arm — All subjects including TB subjects in 5-18 years old、non-TB subjects in 5-18 years old、TB subjects under 5 years old and non-TB subjects under 5 years old inject ESAT6-CFP10 in right arm and TB-PPD in left arm respectively. Two drug must use at the same participant and in different arms.

SUMMARY:
In this clinical research,48 cases TB (Tuberculosis patients) participants and 48 cases non-TB participants with lung disease who all meet the standard are divided into different groups through a randomized and blind method. Every subject inject intradermally ESAT6-CFP10 and TB-PPD (tuberculin purified protein derivative) in different arms of the same person by blind method. Specific gama-interferon (γ-IFN) detection is needed before the injection.Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h. At the same time, we observe all kind of adverse events in order to assess the safety of drug.

DETAILED DESCRIPTION:
In this clinical research,we make sure of the safety in the crowd 5-18 years old firstly,then carry out the crowd of under 5 years old(including 5).

Firstly, 24 cases TB (Tuberculosis) participants and 24 cases non-TB participants with lung disease who are all 5-18 years old and meet the standard respectively are divided into different groups through a randomized and blind method.

1. ESAT6-CFP10(10ug/ml) in left arm and TB-PPD in right arm
2. ESAT6-CFP10(10ug/ml) in right arm and TB-PPD in left arm Inject intradermally ESAT6-CFP10 and TB-PPD in different arms of the same participant. For each of participant, the person in this clinical research, the study uniform is that every subject injects firstly left arm, observe no obvious adverse reaction, then another drug inject in right arm. Measure the induration and (or) redness of longitudinal diameter size and transverse diameter vernier caliper by vernier caliper after injection 24h, 48h and 72h. At the same time, we observe the vital signs (breathing, heart rate, blood pressure and temperature), local reactions (rash, pain, itching and skin mucous membrane) and a variety of adverse events.

Secondly, 24 cases TB (Tuberculosis) participants and 24 cases non-TB participants with lung disease who are all less than 5 years old are divided into two different groups and the procedure are as the same as 5-18 years old.

Finally, we calculate the sensitivity (positive coincidence rate) by TB (Tuberculosis patients), the specificity (negative coincidence rate) by non-TB participants with lung disease, and verify the safety and effectiveness of ESAT6-CFP10(10ug/ml) for the clinical auxiliary diagnosis of tuberculosis.

ELIGIBILITY:
Inclusion Criteria of TB (tuberculosis:include pulmonary tuberculosis and extra pulmonary tuberculosis) subjects:

* judge the pulmonary tuberculosis patient ,according to Chinese Medical Association branch of pediatrics breathing group: Tuberculosis Clinical Diagnostic Criteria and Treatment Programs for Child (trial) ;
* less than 18 years old ,no gender limited;
* Consent and signed informed consent forms (ICF) by the subject or the guardian;
* The subject or with the help of guardian(s) comply with follow-up.

Inclusion Criteria of extra pulmonary tuberculosis subjects:

* Diagnosed extra pulmonary tuberculosis by epidemiology, imaging, clinical symptoms, pathological examination and so on;
* Lesions outside the lungs;
* be in unfinished reinforced phase by chemotherapy;

Exclusion Criteria of TB (tuberculosis) subjects:

* Accompanied by the following severe illness: cancer, acute/progressive liver disease or kidney disease,autoimmune disease，diabetes, primary immunodeficiency diseases, other chronic diseases;
* Taking part in other clinical or within three months involved in any other clinical;
* Severe allergic constitution or familial history of allergy:allergic to two or more drugs;
* in pregnancy or lactation;
* in a mental illness;
* Any conditions affect the trial evaluation by investigator's judgement.

Inclusion Criteria of non-TB participants with lung disease:

* A clear respiratory disease but can exclude pulmonary tuberculosis by clinical symptoms, imaging, laboratory examination.
* less than 18 years old ,no gender limited;
* Consent and signed informed consent forms (ICF) by the subject or the guardian;
* The subject or with the help of guardian(s) comply with follow-up.

Exclusion Criteria of non-TB participants with lung disease:

* Accompanied by the following severe illness: cancer, acute/progressive liver disease or kidney disease,autoimmune disease，diabetes, primary immunodeficiency diseases, other chronic diseases， ect;
* Taking part in other clinical or within three months involved in any other clinical;
* Severe allergic constitution or familial history of allergy: allergic to two or more drugs;
* in pregnancy or lactation;
* in a mental illness;
* active tuberculosis close contactor;
* Any conditions affect the trial evaluation by investigator's judgement.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2016-10; Primary Completion 2017-10 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
The diameter of induration or redness at the injection sites measured transversely to the long axis of the forearm 24 hours、48 hours and 72 hours after application of the agents | From injections to 1-3 days after aplication
  After skin test 1-3d,subjects's injection site may appear inuration or redness .The diameters of induration or redness are measured and recorded.The number of diameter of induration or redness<5mm，the result is negtive.If the number of diameter are not lower than 5mm,the result is positive.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | within 72h after injection two drug each participant
  Any AE of every subject appeared is recorded and traced after signing ICF,until remission of AE.

CONTACTS AND LOCATIONS:
Overall Officials: Shuihua Lu, BBachelor, Principal Investigator — Shanghai Public Health Clinical Center
Locations (4):
- China (4):
  - Wuhan Medical Treatment Center, Wuhan, Hubei
  - Beijing Children's Hospital, Beijing
  - Shanghai Public Health Clinical Center, Shanghai
  - Wuhan Institute for Tuberculosis Control, Wuhan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Pinxteren LA, Ravn P, Agger EM, Pollock J, Andersen P. Diagnosis of tuberculosis based on the two specific antigens ESAT-6 and CFP10. Clin Diagn Lab Immunol. 2000 Mar;7(2):155-60. doi: 10.1128/CDLI.7.2.155-160.2000. PMID 10702486
- [Background] Brusasca PN, Colangeli R, Lyashchenko KP, Zhao X, Vogelstein M, Spencer JS, McMurray DN, Gennaro ML. Immunological characterization of antigens encoded by the RD1 region of the Mycobacterium tuberculosis genome. Scand J Immunol. 2001 Nov;54(5):448-52. doi: 10.1046/j.1365-3083.2001.00975.x. PMID 11696195
- [Background] Weldingh K, Andersen P. ESAT-6/CFP10 skin test predicts disease in M. tuberculosis-infected guinea pigs. PLoS One. 2008 Apr 23;3(4):e1978. doi: 10.1371/journal.pone.0001978. PMID 18431468
- [Background] Aagaard C, Govaerts M, Meikle V, Vallecillo AJ, Gutierrez-Pabello JA, Suarez-Guemes F, McNair J, Cataldi A, Espitia C, Andersen P, Pollock JM. Optimizing antigen cocktails for detection of Mycobacterium bovis in herds with different prevalences of bovine tuberculosis: ESAT6-CFP10 mixture shows optimal sensitivity and specificity. J Clin Microbiol. 2006 Dec;44(12):4326-35. doi: 10.1128/JCM.01184-06. Epub 2006 Sep 27. PMID 17005738